CLINICAL TRIAL: NCT04743310
Title: A Phase 2 Study of Fluorescence Detection of Adult Primary Central Nervous System Tumors in Subjects Receiving Tozuleristide and Imaged With the Canvas System
Brief Title: Fluorescence Detection of Adult Primary Central Nervous System Tumors With Tozuleristide and the Canvas System
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: John Yu (Other)
Collaborators: Blaze Bioscience Inc. (Industry)
Responsible Party: Sponsor-Investigator, John Yu, Director, Surgical Neuro-Oncology, Cedars-Sinai Medical Center
Organization: Cedars-Sinai Medical Center (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IIT2020-09-Yu-BBIST001
Record Dates: First submitted 2021-02-04; First posted 2021-02-08 (Actual); Last update posted 2025-06-13 (Actual); Status verified 2025-06

CONDITIONS: Central Nervous System Tumor
Keywords: neurosurgery; brain tumor; spinal cord tumor; surgical resection; glioma; astrocytoma; glioblastoma; ependymoma; medulloblastoma; pineocytoma; meningioma; germ cell tumor; craniopharyngioma; oligoastrocytoma; pineoblastoma; extent of resection; maximal safe resection; neuropathology; vestibular schwannomas
MeSH Terms: conditions — Central Nervous System Neoplasms; Brain Neoplasms; Spinal Cord Neoplasms; Glioma; Astrocytoma; Glioblastoma; Ependymoma; Medulloblastoma; Pinealoma; Meningioma; Neoplasms, Germ Cell and Embryonal; Craniopharyngioma; Neuroma, Acoustic | interventions — tozuleristide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (1):
- Tozuleristide with Canvas imaging system (Experimental)
  Interventions: Drug: tozuleristide; Device: Canvas imaging system; Procedure: Surgical resection of tumor

INTERVENTIONS:
Drug: tozuleristide — tozuleristide 24 or 36 mg administered intravenously 1-24 hours prior to surgery
Device: Canvas imaging system — imaging device attached to surgical microscope
Procedure: Surgical resection of tumor — Standard of care surgical resection of tumor

SUMMARY:
The purpose of this study is to examine the use of a single dose of tozuleristide (24 or 36 mg) and the Canvas imaging system during surgical resection of primary central nervous system (CNS) tumors: Primary gadolinium enhancing (high grade) CNS tumors, primary non-gadolinium enhancing CNS tumors, and primary vestibular schwannoma.

The primary objectives of the study is to see how well tozuleristide and the Canvas imaging system during surgical resection will show fluorescence among primary enhancing/high grade CNS tumors; and among the tumors that demonstrate tozuleristide fluorescence, to estimate the true positive rate and true negative rate of fluorescence in tissue biopsies, as well as sensitivity and specificity of tozuleristide fluorescence for distinguishing tumor from non-tumoral tissue.

The secondary objectives of the study include evaluating the safety of tozuleristide and the Canvas imaging system, and to determine if the presence of remaining fluorescence at the time of surgery corresponds to remaining tumor evident on post-operative MRI images, or if the absence of fluorescence corresponds to evidence of no gross residual tumor on post-operative magnetic resonance imaging (MRI).

ELIGIBILITY:
Inclusion Criteria:

* MRI obtained within 30 days of study enrollment documents a measurable lesion consistent with a primary malignant central nervous system tumor for which maximal safe resection is indicated OR MRI obtained within 30 days of study enrollment documents a measurable lesion consistent with a primary schwannoma enhancing tumor in the cerebellopontine angle for which maximal safe resection is indicated.
* Adequate renal and liver function
* Subjects with prior therapy are eligible provided they have recovered from any acute toxic effects of prior therapy and have sufficient time interval prior to enrollment.

Exclusion Criteria:

* Pregnant, breast-feeding, or planning to conceive a child within 30 days
* Ongoing serious medical conditions such that participation in the study could put the subject at increased risk of worsening their condition
* Subjects planned to undergo only a diagnostic biopsy procedure, without intent to resect tissue for therapeutic purposes
* Subjects for whom radiographic evidence suggests a non-intra-axial primary brain tumor

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2021-09-30 (Actual); Primary Completion 2025-03-06 (Actual); Study Completion 2025-03-06 (Actual)

PRIMARY OUTCOMES:
Percentage of patients with fluorescence-positive primary tumor biopsy | At the time of surgery
True positive rate of fluorescence, defined as the percentage of tumor-positive and fluorescence-positive tissue biopsies among all tumor-positive tissue biopsies | At the time of surgery
True negative rate of fluorescence, defined as the percentage of tumor-negative and fluorescence-negative tissue biopsies among all tumor-negative tissue biopsies | At the time of surgery

SECONDARY OUTCOMES:
Positive predictive value of fluorescence, defined as the percentage of tumor-positive and fluorescence-positive tissue biopsies among all fluorescence-positive tissue biopsies | At the time of surgery
Negative predictive value of fluorescence, defined as the percentage of tumor-negative and fluorescence-negative tissue biopsies among all fluorescence-negative tissue biopsies | At the time of surgery
Extent of residual tumor measured on post-operative magnetic resonance imaging scans among all patients with evidence of residual fluorescence at the time of surgery | At the time of surgery

OTHER OUTCOMES:
Incidence of adverse events | From the time of study drug administration 1-24 hours prior to surgery, until 30 days after surgery or until receiving additional therapy for the central nervous system tumor, whichever comes first
  Recorded and graded according to the National Cancer Institute's Common Terminology Criteria for Adverse Events Version 5

CONTACTS AND LOCATIONS:
Overall Officials: John Yu, MD, Principal Investigator — Cedars-Sinai Medical Center
Locations (1):
- Cedars-Sinai Medical Center, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: No